CLINICAL TRIAL: NCT02230241
Title: CEntralized Pan-Russian Survey of tHE Undertreatment of hypercholeSterolemia II
Brief Title: CEntralized Pan-Russian Survey of tHE Undertreatment of hypercholeSterolemia II (CEPHEUS II)
Acronym: CEPHEUSII
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-CRU-XXX-2014/1
Record Dates: First submitted 2014-08-26; First posted 2014-09-03 (Estimated); Last update posted 2016-05-05 (Estimated); Status verified 2016-05

CONDITIONS: Dyslipidaemia
Keywords: Dyslipidaemia; LDL-C goals; Guidelines
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cohort 1: Subjects of either gender and any race, aged ≥ 18 years, at moderate to very high CV risk, on lipid-lowering pharmacotherapy for at least 3 months (90 days), with no dose change for a minimum of 8 weeks (56 days). Before starting any study-related activities, the investigator should obtain written informed consent personally signed and dated by the subject.

SUMMARY:
This is a multi-center survey of patients who are currently receiving lipid-lowering medications and have a moderate or higher cardiovascular (CV) risk. The survey will be conducted in the Russian Federation. Data collection for each study subject will be done within one physician visit. If an enrolled subject comes to the visit not fasting (for at least 8 hours), an appointment for the blood tests will be made for another day.

DETAILED DESCRIPTION:
This is a multi-center survey of patients who are currently receiving lipid-lowering medications and have a moderate or higher CV risk. The survey will be conducted in the Russian Federation.

Data collection for each study subject will be done within one physician visit. If an enrolled subject comes to the visit not fasting (for at least 8 hours), an appointment for the blood tests will be made for another day.

Prior to the assessment of the first subject at a site, each investigator will complete an investigator questionnaire on his/her experience and perception of the management of hypercholesterolemia in his/her patients.

Prior to the assessment, subjects will record on a patient questionnaire their awareness of hypercholesterolemia, their current treatment schedule, their perception, and compliance.

The investigator will complete a Case Report Form (CRF) with the subject's demographics, known cardiovascular risk factors, cardiovascular medical history, current lipid-lowering drug therapy, and the reason for this therapy.

Fasting blood samples will be taken in tubes to test for total cholesterol, low-density lipoprotein cholesterol (LDL), high-density lipoprotein cholesterol (HDL), glucose, creatinine, hemoglobin A1c, hemoglobin, and hematocrit at a central laboratory in the Russian Federation.

ELIGIBILITY:
Inclusion Criteria:

* Properly obtained written informed consent from the potential subject.
* On lipid-lowering drug therapy for at least 3 months (90 days), with no dose change for a minimum of 8 weeks (56 days).
* Scheduled blood tests for total cholesterol (TC), HDL-C, LDL-C, glucose, creatinine, HbA1c, Hb, and hematocrit on the visit when they are considered for survey participation, or these tests must be decided to be necessary for study-unrelated purposes during that visit.

Exclusion Criteria:

* Subjects who are unwilling or unable to provide written informed consent.
* The cognitive status of a potential subject and/or their home environment (in the investigator's opinion) might compromise the compliance with the treatment regimen during the past 8 weeks.
* A low CV risk.
* Participating in any other clinical trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects of either gender and any race, aged ≥ 18 years, at moderate to very high CV risk, on lipid-lowering pharmacotherapy for at least 3 months (90 days), with no dose change for a minimum of 8 weeks (56 days). Before starting any study-related activities, the investigator should obtain written informed consent personally signed and dated by the subject.
Sampling Method: Non-Probability Sample
Enrollment: 2700 (Actual)
Dates: Start 2014-09; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
The proportion of patients who reach the low-density lipoprotein cholesterol (LDL-C) goals established by the Fifth Joint European Task Force guidelines (2012). | Up to 11 months

SECONDARY OUTCOMES:
The proportion of patients at moderate to very high CV risk on lipid-lowering drug therapy who reach the LDL-C goals per the Fifth Joint European Task Force guidelines in the following sub-populations | Up to 11 months
The percentage of incorrect CV-risk assessments made by physicians | Up to 11 months
The proportion of subjects in a subgroup of those with diabetes mellitus and interpretable Hemoglobin A1c (HbA1c) results who achieve HbA1c standardized target of 7% (per Diabetes Control and Complications Trial - DCCT1). | Up to 11 months

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Bedenkov, Study Director — AstraZeneca; Sergey Boytsov, Principal Investigator — State Research Center for Preventive Medicine MoH
Locations (27):
- Russia (27):
  - Research Site, Belgorod
  - Research Site, Berdsk
  - Research Site, Domodedovo
  - Research Site, Engel's
  - Research Site, Ivanovo
  - Research Site, Kaluga
  - Research Site, Kirovsk
  - Research Site, Korolyov
  - Research Site, Krasnodar
  - Research Site, Krasnoyarsk
  - Research Site, Moscow
  - Research Site, Mytishchy
  - Research Site, Nizhny Novgorod
  - Research Site, Novosibirsk
  - Research Site, Odintsovo
  - Research Site, Orenburg
  - Research Site, Penza
  - Research Site, Pushkino
  - Research Site, Rostov-on-Don
  - Research Site, Saint Petersburg
  - Research Site, Samara
  - Research Site, Sergiyev Posad
  - Research Site, Sochi
  - Research Site, Volgograd
  - Research Site, Voronezh
  - Research Site, Yaroslavl
  - Research Site, Yekaterinburg

REFERENCES:
- [Derived] Boytsov S, Logunova N, Khomitskaya Y; CEPHEUS II investigators. Suboptimal control of lipid levels: results from the non-interventional Centralized Pan-Russian Survey of the Undertreatment of Hypercholesterolemia II (CEPHEUS II). Cardiovasc Diabetol. 2017 Dec 16;16(1):158. doi: 10.1186/s12933-017-0641-4. PMID 29246151
- See also: Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3105&filename=CEPHEUSII_NISPrimaryReport_Synopsis.pdf